CLINICAL TRIAL: NCT06285708
Title: Enhancing the Effectiveness of Prolonged Exposure Among Suicidal Individuals With PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023B0193
Record Dates: First submitted 2024-02-14; First posted 2024-02-29 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: PTSD; Suicidal Ideation; Suicide, Attempted; Trauma, Psychological
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation; Suicide, Attempted; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged exposure with crisis response plan (Experimental): In the enhanced prolonged exposure condition, participants will complete a CRP instead of a safety plan. The CRP is another recommended standard care practice with suicidal patients that includes many of the same elements as the safety plan (i.e., warning signs, self-management strategies, sources of social support, crisis services), but is created collaboratively by the patient with active input of their clinician rather than being self-guided. The CRP also includes a section focused on the participant's reasons for living, an addition that has been shown to increase positive emotional states (e.g., hope, optimism) and lead to faster reductions in suicidal intent. The CRP will be administered during the first therapy session.
  Interventions: Behavioral: Prolonged exposure
- Prolonged exposure with safety plan (Active Comparator): In the standard prolonged exposure condition, participants will complete a safety plan, a procedure that includes personal warning signs for a suicidal crisis, self-management strategies, sources of social support, and contact information for professional resources and crisis services within the participant's local community, as well as the National Suicide Prevention Lifeline phone number. As a recommended standard care practice with suicidal patients, the combination of PE and safety plan represents treatment as usual. The safety plan will be administered during the first therapy session.
  Interventions: Behavioral: Prolonged exposure

INTERVENTIONS:
Behavioral: Prolonged exposure — PE therapy is a manualized cognitive behavioral therapy consisting of imaginal exposure (repeated recounting of the most disturbing traumatic memory) followed by processing thoughts and feelings related to the imaginal experience; in-vivo exposure (approaching trauma-related situations); psychoeducation about PTSD; and controlled breathing training. Between sessions, participants listen to audio recordings of the imaginal recounting daily and complete in-vivo exercises. Typically, PE is delivered weekly for 10-12, 90-minutes sessions. For this study, participants will complete daily 60-minute sessions for 10 consecutive weekdays during a 2-week period.

SUMMARY:
The long-term goal of this study is to reduce suicidal thoughts and behaviors among treatment-seeking individuals who also have posttraumatic stress disorder (PTSD). Prolonged exposure (PE) and crisis response plan (CRP) have demonstrated empirical support for reducing suicide attempts as compared to treatment as usual. However, no studies to date have assessed their effectiveness when used in combination. In light of this knowledge gap, the primary objective of this study will be to test the effectiveness of PE augmented with CRP as compared to PE with care as usual (self-guided treatment plan), an active comparator, for the reduction of suicide ideations and attempts for individuals with comorbid PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is associated with a host of functional problems and negative outcomes, including occupational and marital dissatisfaction, violence, alcohol and substance abuse, and suicide. Cognitive behavioral treatments tend to be the most highly efficacious treatments for PTSD. Prolonged Exposure (PE) therapy is a manualized cognitive behavioral therapy consisting of imaginal exposure followed by processing thoughts and feelings related to the imaginal experience; in-vivo exposure, psychoeducation, and controlled breathing training. Preliminary evidence suggests that PE is associated with significant suicidal ideation (SI) reductions. Enhancing PE with procedures that have been shown to significantly reduce suicidal thoughts and behaviors could serve to further reduce suicide risk during and after treatment completion.

The long-term goal of this project is to prevent suicides among individuals diagnosed with PTSD by integrating trauma-focused therapies with suicide-focused interventions. The primary objective of this pilot project is to test the efficacy of PE when enhanced with a crisis response plan utilizing self-report, behavioral, and ecological assessment methods to compare treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of PTSD or subthreshold PTSD; ability to speak and understand the English language; and ability to complete the informed consent process.

Exclusion Criteria:

* Substance use disorder requiring medical management; imminent suicide risk warranting inpatient hospitalization or suicide-focused treatment; and impaired mental status that precludes the ability to provide informed consent (e.g., intoxication, psychosis, mania).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Beck Scale for Suicidal Ideation (SSI) | During the first 3 weeks and through one year follow up
  19 item self-report assessment of suicidal ideation, range of scores is 0-57, higher score indicates higher suicidal ideation
Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R) | During the first 3 weeks and through one year follow up
  31 item self-report measure of suicidal thoughts and behavior
PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (PCL-5) | During the first 3 weeks and through one year follow up
  20 item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. range is 0-80, higher score indicates higher PTSD symptoms

SECONDARY OUTCOMES:
Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Self-Rated Level 1 Cross-Cutting Symptom Measure | During the first 3 weeks and through one year follow up
  transdiagnostic measure of current mental health symptomatology. It is an adult measure that consists of 23 questions that assess 13 psychiatric domains, including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use.
Interpersonal Needs Questionnaire (INQ) - Abbreviated | During the first 3 weeks and through one year follow up
  self-report assessment of interpersonal factors (perceived burdensomeness and thwarted belongingness) that contribute to suicidal ideation.
Beck Hopelessness Scale (BHS) - Abbreviated | During the first 3 weeks and through one year follow up
  A 5 item self-report assessment of hopelessness, range of scores is 0-10, higher scores indicate better outcome
Brief Suicide Cognitions Scale (SCS) | During the first 3 weeks and through one year follow up
  6 item self-report assessment of thoughts related to suicidal ideation, range of scores is 0-30, higher score indicates worse outcome
Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) | During the first 3 weeks and through one year follow up
  self-report assessment of emotion regulation.
Monetary Choice Questionnaire (MCQ) | During the first 3 weeks and through one year follow up
  a self-report assessment of impulsivity
Behavioral Inhibition Scale (BIS) | During the first 3 weeks and through one year follow up
  a 7 item self-report assessment of punishment sensitivity, range 0-28, higher scores indicate worse outcome
Behavioral Activation Scale (BAS) | During the first 3 weeks and through one year follow up
  a 13 item self-report assessment of reward sensitivity, range 0-52, higher scores indicate worse outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures | During the first 3 weeks and through one year follow up
  a 4 item self-report assessment of depression, range of scores 4-20, higher score indicates worse outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures | During the first 3 weeks and through one year follow up
  a 4 item self-report assessment of anxiety, range of scores 4-20, higher scores indicate worse outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures | During the first 3 weeks and through one year follow up
  a 4 item self-report assessment of social activity, range of scores is 4-20, higher score indicates worse outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures | During the first 3 weeks and through one year follow up
  a 4 item self-report assessment of fatigue, range of scores is 4-20, higher scores indicate worse outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures | During the first 3 weeks and through one year follow up
  a 4 item self-report assessment of sleep, range of scores is 4-20, higher scores indicate worse outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures | During the first 3 weeks and through one year follow up
  a 4 item self-report assessment of physical function, range of scores is 4-20, higher score indicates better outcome
Patient-Reported Outcomes Measurement Information System (PROMIS) Measures | During the first 3 weeks and through one year follow up
  a 5 item self-report assessment of pain, range of scores 5-25, higher scores indicates worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jaryd Hiser, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data available by request